CLINICAL TRIAL: NCT06204068
Title: A Prospective Analysis of Optimal Spica Cast Duration Following Closed Reduction for Developmental Dysplasia of the Hip (DDH)
Brief Title: Spica Cast Duration for DDH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrolment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000035569; 000 (Other: CTGTY)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Dysplasia; Hip
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hip Spica 6 weeks, Brace 6 weeks (Experimental): The experimental group will be placed in a hip spica cast for a total of 6 weeks, then will transition to a brace for 6 weeks.
  Interventions: Device: Spica cast; Device: Rhino brace
- Hip Spica 12 weeks (Control) (Active Comparator): The control group will be placed in a hip spica cast for a total of 12 weeks with a change of spica cast, under anesthesia, at the 6-week mark. This treatment is the accepted standard of care for children who undergo closed reduction of a developmentally dysplastic and dislocated hip.
  Interventions: Device: Spica cast

INTERVENTIONS:
Device: Spica cast — Spica cast is a cast that is placed while the child is sedated or under anesthesia, covering lower part of belly, waist, and both legs made up of fiberglass, also keeps legs in abduction and flexion. This device will be used as intended and is commonly used for the treatment of DDH.
Device: Rhino brace — Hip abduction brace will be used, which keeps the legs abducted and flexed. A hip brace is a special type of brace that is designed to hold the hips in a flexed and abducted position. This position allows the hip joint to develop properly while it heals. This device will be used as intended and is commonly used for the treatment of DDH.
  Arms: Hip Spica 6 weeks, Brace 6 weeks

SUMMARY:
This study looks at treatment for developmental dysplasia of the hip (DDH), a condition where there is abnormal development of a child's hip joint. While spica casts are shown to very effective in treating DDH, and potentially more effective than hip braces alone, other research shows that the outcomes from braces are equivalent to those of spica casts with the added advantage of greater patient satisfaction and less burden on families. Therefore, the 12-week experimental protocol in the study, with the first 6 weeks involving the spica cast and the second 6 weeks the hip brace, was designed to determine if both treatment methods can be combined for an optimal patient experience.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the clinical outcomes of patients who undergo closed reduction of a developmentally dysplastic hip and are treated with six weeks of supplemental casting to those treated with twelve weeks of supplemental casting.

The secondary objectives of this study are to determine if a shorter duration of postoperative casting affects family satisfaction and costs compared to the traditional pathway (12 weeks of spica casting).

The physician will meet with the patients during the regular standard of care follow-ups every 2-3 weeks to track patient progress. Following 6 weeks of recovery, the control group will have their spica cast replaced in the operating room, with the child anesthetized, by another cast for 6 weeks. The experimental group will have their cast removed in the clinic without anesthesia and will be placed into a full-time brace for 6 weeks. Participants will be instructed to complete the full 12 weeks of the protocols. Only patients who complete the full length of treatment in either group will be considered for the study. The physicians will keep track of patients during visits to ensure the protocols are being followed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with DDH
* Require closed reduction of the hip and hip spica casting

  1. between 6-18 months old
  2. Alpha angle <60 degrees, beta angle >55 degrees

  i. Alpha angle is an angle created by lines along bony acetabulum and the ilium, normal is >60 degrees

ii. Beta angle is an angle created by lines along the labrum and ilium, normal is <55 degrees

c.Have either failed Pavlik harness or have dislocated hip on imaging

Exclusion Criteria:

* Patients over the age of 18 months
* Patients with DDH who do not require closed reduction surgery
* Patients with DDH who are initially consented for closed reduction surgery but their intraoperative findings necessitate conversion to open surgery
* Families that do not want to participate in the study
* Patients with dysplasia that need open reduction

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Re-Dislocation Rate | up to 12 weeks
  The incidence of DDH re-occurrence in patients over the 12 week course of the casting or bracing for early re-dislocation rate. This will be the main quantitative value that directly measures the effectiveness of the protocols on maintaining the results of the closed reduction surgery.
Patient Satisfaction Scores using Pediatric Outcome Questionnaire | 6 weeks and 12 weeks
  Pediatric Outcome Questionnaire - 86 questions, item scores are summed for a total score. Total score range from 0-100, Higher score means higher satisfaction.
Complications Rate | up to 12 weeks
  The incidence of any complications that occur over the 12 week course.
Hospital Re-Admission Rate | up to 12 weeks
  Number of participants re-admitted to the hospital
Mean Time to Hospital Re-Admission | up to 12 weeks
  Mean Time to Hospital Re-Admission in days

SECONDARY OUTCOMES:
Family Satisfaction/Burden using Pediatric Outcome Questionnaire | 12 weeks
  Pediatric Outcome Questionnaire - 86 questions, item scores are summed for a total score. Total score range from 0-100, Higher score means higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Tuason, MD, Principal Investigator — Yale University; Adrienne Socci, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No